CLINICAL TRIAL: NCT01806077
Title: Demonstration of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Antiplatelet Effect of PZ-128 in Subjects With Multiple Coronary Artery Disease Risk Factors
Brief Title: Safety Study of PZ-128 in Subjects With Multiple Coronary Artery Disease Risk Factors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Sinai Hospital of Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TMC-A2012-04; P50HL110789 (NIH)
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Vascular Disease; Coronary Artery Disease Risk Factors Multiple
Keywords: Cardiovascular Diseases; Vascular Diseases; Coronary Artery Disease; Coronary Disease; Arteriosclerosis; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Vascular Diseases; Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Arteriosclerosis | interventions — PZ-128 peptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PZ-128 (Experimental)
  Interventions: Drug: PZ-128

INTERVENTIONS:
Drug: PZ-128 — Sequential single-dose escalation; 1 to 2 hour continuous intravenous infusion

SUMMARY:
This study is a Phase I, intravenous, single-dose escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of PZ-128 (pepducin inhibitor of PAR1) in subjects with vascular disease or who have 2 or more coronary artery disease (CAD) risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 75 with documented vascular disease (peripheral vascular disease, carotid artery disease or coronary artery disease) or 2 or more coronary artery risk factors.
* Women of childbearing potential must have a negative pregnancy test prior to enrollment and immediately before drug administration and agree to use two methods of effective barrier contraception, or a hormonal contraceptive to prevent pregnancy throughout the study.
* The subject is able to read and give written informed consent and has signed and dated an informed consent document and authorization permitting release of personal health information approved by the Investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* The subject has participated in an investigational drug study within the last 30 days.
* The subject has a medical or surgical condition that may impair drug absorption or metabolism.
* Anticoagulants, P2Y12 inhibitors, nonsteroidal antiinflammatory drugs (no more than three times a week) or any other drug that the investigator deems to have potential interaction with platelets or PAR-1 receptor inhibition are prohibited from 2 weeks prior to study drug dosing through 2 weeks post dosing. Aspirin is allowed.
* The subject has previous history of anaphylaxis to drugs or any environmental stimuli including foods or hymenoptera (e.g., ants, bees, wasps) stings.
* Asthma requiring bronchodilator/inhaler therapy.
* Currently smoking ≥2 pack/day.
* Herbal supplements (i.e., Fish Oil/Omega-3, St. John's Wart, Ginseng, Garlic, Ginkgo, Saw Palmetto, Echinacea, Yohimbine, Licorice, and Black Cohosh) are prohibited from 1 week prior to dosing through 24 hours post dosing.
* Prior history or clinical suspicion of cerebral vascular malformations, intracranial tumor, transient ischemic attack, stroke, gastric ulcers and any form of bleeding disorder.
* Prior history of myocardial infarction within the last 3 months or unstable angina.
* Thrombocytopenia defined as a platelet count of <130,000/mm3 or low hematocrit defined as <30%.
* Renal function: serum creatinine >1.5 x ULN. However, subjects with an estimated creatinine clearance eGFR ≥60 mL/min, calculated using the Cockcroft-Gault formula, are eligible.
* Liver enzymes ≥ 3 x upper limit of normal.
* Alcohol consumption within 48 hrs prior to dosing, and for the duration of the in-house study period.
* Evidence of history of substance or alcohol abuse at screening, including positive urine test results for drugs or positive breath test for alcohol.
* Uncontrolled hypertension or hypotension defined as a sustained supine systolic pressure >160 mmHg or <100 mmHg; or a diastolic pressure >90 mmHg or < 50 mmHg.
* International normalized ratio (INR) >1.5
* Poor venous access (i.e., insufficient for intravenous drug delivery).
* History of hepatitis or HIV.
* The subject has undergone an invasive surgical procedure within the last 3 months, is anticipating one during the course of their study participation or is planning to have one within 1 month post dosing with the study drug.
* The subject has any condition which could interfere with or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the Investigator increase the risk of the subject's participation in the study. This would include, but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy or any unexplained blackouts, previous hypersensitivity to drugs, and severe asthma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Summary of Participants Experience with Safety and Tolerability | 30 days after drug infusion
  Safety and tolerability of a single dose of PZ-128 as determined by adverse event reporting, clinical laboratory results, vital signs, physical examination, pulmonary function tests and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Pharmacokinetic profile of PZ-128 | Assessments will be done up to 7 days post dosing
Evaluate inhibition of ex vivo platelet function in response to multiple agonists | Assessments will be done up to 7 days post dosing
Correlate PZ-128 plasma levels with inhibition of platelet aggregation | Assessments will be done up to 7 days post dosing
Evaluate changes in clotting characteristics at each dose level of PZ-128 relative to baseline | Assessments will be done up to 7 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Gurbel, MD, Principal Investigator — Sinai Hospital of Baltimore (Sinai Center for Thrombosis Research); Athan Kuliopulos, MD, PhD, Study Director — Tufts Medical Center (Hemostasis and Thrombosis Laboratory)
Locations (1):
- Sinai Hospital of Baltimore (Sinai Center for Thrombosis Research), Baltimore, Maryland, United States

REFERENCES:
- [Background] Gurbel PA, Bliden KP, Turner SE, Tantry US, Gesheff MG, Barr TP, Covic L, Kuliopulos A. Cell-Penetrating Pepducin Therapy Targeting PAR1 in Subjects With Coronary Artery Disease. Arterioscler Thromb Vasc Biol. 2016 Jan;36(1):189-97. doi: 10.1161/ATVBAHA.115.306777. PMID 26681756